CLINICAL TRIAL: NCT06120166
Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10- 19) in the Treatment of r/r DLBCL Clinical Research
Brief Title: Safety and Efficacy of Metabolically Armed CD19 CAR-T Cells (Meta10-19) in the Treatment of r/r DLBCL Clinical Research
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: He Huang (Other)
Collaborators: Leman Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, He Huang, Clinical Professor, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Meta10-19-003
Record Dates: First submitted 2023-10-25; First posted 2023-11-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Meta10-19; CAR-T Cells Therapy; r/r DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Administration of Metabolically Armed CD19 CAR-T cells (Experimental): Patients undergo leukapheresis. Patients will receive a lymphodepletion chemotherapy with cyclophosphamide and fludarabine before CAR-T cells infusion. A dose of metabolically armed CD19 CAR-T cells will be infused on day 0.
  Interventions: Drug: Metabolically Armed CD19 CAR-T cells

INTERVENTIONS:
Drug: Metabolically Armed CD19 CAR-T cells — Each subject receive metabolically armed CD19 CAR-T cells by intravenous infusion
  Other Names: Meta10-19

SUMMARY:
A Study of Metabolically Armed CD19 CAR-T Cells Therapy for Patients With Relapsed and/or Refractory Diffuse Large B-Cell Lymphoma

DETAILED DESCRIPTION:
This is a single arm, open-label study. This study is indicated for relapsed or refractory CD19+ Diffuse Large B-Cell Lymphoma. The selections of dose levels and the number of subjects are based on clinical trials of similar foreign products.

1. Main research objectives:

   To evaluate the safety and efficacy of metabolically armed CD19 CAR-T Cells in the treatment of r/r DLBCL.
2. Secondary research objectives:

   1. To evaluate the pharmacokinetic (PK) and pharmacodynamics(PD) characteristics of metabolically armed CD19 CAR-T Cells after infusion.
   2. To evaluate tumor remission after infusion of metabolically armed CD19 CAR-T Cells.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her guardian voluntarily signed the informed consent
* Adult Patients clinical diagnosis of relapsed and refractory diffuse large B-cell lymphoma (Primary mediastinal large B-cell lymphoma and transformed follicular lymphoma are included)

Definition of refractory:

1. No response to the last treatment, including:

   The best response to the last treatment was PD, or ; The best response to the last treatment was SD and the duration was not more than 6 months after the last dose.
2. Not suitable for autologous hematopoietic stem cell transplantation (ASCT), or ASCT refractory, including:

Disease progression or recurrence within 12 months or less (recurrence must be confirmed by biopsy) after ASCT treatment, or; Patients accept remedial treatment after ASCT must have no response or relapse after the last treatment

* Patients who had previously received ≥2 lines therapy including at least:

  1. A chemotherapy regimen containing anthracyclines
  2. For patients with transformed DLBCL from follicular lymphoma, they must have previously received chemotherapy for follicular lymphoma and have refractory disease after transformation to DLBCL.
* Patients with double-strike and triple-strike lymphoma who do not respond to second-line treatment, where double-strike/triple-strike is defined as:

Detection of lymphoma cells with C-MYC gene translocation accompanied by BCL-2 gene translocation or/and BCL-6 gene translocation by chromosome or FISH technology.

* CD19 expression was positive by immunohistochemistry or flow cytometry (accept the results of this peripheral blood mononuclear cells or previous report from a Class A tertiary hospital before peripheral blood collection)
* At least one measurable lesion at baseline, according to the initial assessment, staging and Response Assessment recommendations for Hodgkin's and non-Hodgkin's lymphoma (2014 edition)
* Expected survival time greater than 12 weeks
* The baseline ECOG score was 0 or 1
* Organ function:

  1. Kidney function is defined as:

     Serum creatinine ≤1.5 times ULN, or; The glomerular filtration rate (eGFR) estimated by MDRD formula was ≥60m/ min/1.73m2; [eGFR=186×(age)-0.203×SCr- 1. 154(mg/dl), for females, the result was ×0.742]
  2. Liver function is defined as:

     ALT≤5 times ULN, and; Patients with total bilirubin ≤2.0mg/dl, except those with Gilbert-Meulengracht syndrome. Patients with Gilbert-Meulengracht syndrome with total bilirubin ≤3.0 times ULN and direct bilirubin ≤1.5 times ULN were included
  3. Pulmonary function: ≤CTCAE grade 1 dyspnea and oxygen saturation of blood (SaO2) ≥91% in indoor air environment.
* Hemodynamic stability was determined by echocardiography or multichannel radionuclide angiography (MUGA) and LVEF ≥45%
* Patients using the following drugs must meet the following conditions:

  1. Steroid: Therapeutic doses of steroids must be discontinued 2 weeks prior to Meta10-19 infusion. However, physiological replacement doses of steroids are permitted, hydrocortisone or its equivalent <6-12mg/mm2/ day
  2. Immunosuppressive agent: Any immunosuppressive drug must be stopped ≥4 weeks before the informed consent is signed
  3. Anti-proliferative therapy in addition to preconditioning chemotherapy 2 weeks prior to Meta10-19 infusion
  4. Treatment for CNS disease must be stopped 1 week before Meta10- 19 infusion (e.g., intrathecal methotrexate)
* The patient has recovered from the toxicity of the previous treatment, that is, the CTCAE toxicity grade is less than 1 (The exception is specific toxicity of grade 2 or less, such as hair loss, which the researchers have determined is not recoverable in a short period of time) is suitable for pretreatment chemotherapy and CAR T cell therapy
* Women of childbearing age and all male patients must consent to use a effective contraception for at least 12 months after Meta10-19 infusion and until two consecutive PCR tests show no more CAR T cells in vivo

Exclusion Criteria:

* Patients with present or history of central nervous system diseases such as seizures disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement
* Patients with history of allogeneic hematopoietic stem cell transplantation
* Patients who had received chemotherapy other than preconditioning chemotherapy within 2 weeks prior to Meta10-19 infusion
* Patients who participated in other clinical trials within 30 days prior to enrollment
* Patients with active hepatitis B (defined as hepatitis B surface antigen positive or hepatitis B core antibody positive, concomitant hepatitis B virus DNA level >1000 copies/ml) or hepatitis C (HCV RNA positive)
* Patients with HIV antibody positive or treponema pallidum antibody positive
* Patients with uncontrolled acute life-threatening bacterial, viral or fungal infections (e.g. positive blood cultures ≤72 hours before Meta10-19infusion)
* Patients with unstable angina pectoris and/or myocardial infarction within 6 months prior to enrollment
* Patients with history of other malignancies, but the following conditions can be enrollment:

  1. Adequately treated basal or squamous cell carcinoma (requiring adequate wound healing before signing informed consent);
  2. Carcinoma in situ (DCIS) of cervical or breast cancer, which has been treated therapeutically, has shown no signs of recurrence for at least 3 years prior to the signing of the informed consent
  3. The primary malignancy has been completely resected and in complete remission for ≥5 years
* Women who are pregnant or breastfeeding (pregnancy tests for women of childbearing age are positive)
* Patients with active neuroautoimmune or inflammatory conditions (e.g. Guillian-Barre syndrome, amyotrophic lateral sclerosis);
* Other conditions that the investigator considered should not be enrolled in this clinical study, such as poor compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
MTD | MTD will be determined based on DLTs observed during the first 28 days of study treatment.
  Determine the Maximal Tolerable Dose(MTD)
Objective response rate (ORR) | Within 3 months following infusion of Meta10-19
  Measure Tumor response rate (including CR and PR)

SECONDARY OUTCOMES:
Concentration of CAR-T cells | Up to 12 months after CAR-T treatment
  Concentration of CAR-T cells measured by Flow cytometry after CAR-T infusion
Pharmacodynamics of CAR-T cells | Up to 28 days after infusion
  Concentration levels of CAR-T related serum cytokines such as CRP, IL-6, INF-γ at each time point

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No